CLINICAL TRIAL: NCT01986517
Title: Impact of Feedback on the Devolpment of Psychotherapeutic Competencies: a Randomized Controlled Trial
Brief Title: Feedback and Psychotherapeutic Competencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Florian Weck, PhD, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Feedback-01
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Mental Disorders
Keywords: Feedback; Therapeutic competencies; Training
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Experimental): Therapists assigned to this group will receive standardized feedback on their psychotherapeutic competency after every fourth treatment session with a patient for a period of 20 therapy sessions. The feedback will be given by two experienced raters who are licensed as psychological psychotherapists.
  Interventions: Behavioral: Feedback after every fourth session
- No feedback (Experimental): Therapists assigned to this group will receive no feedback
  Interventions: Behavioral: No feedback

INTERVENTIONS:
Behavioral: No feedback — Therapists will receive no feedback.
  Arms: No feedback
Behavioral: Feedback after every fourth session
  Arms: Feedback

SUMMARY:
The purpose of the current study is to examine the influence of feedback on psychotherapeutic competency. The present randomized controlled study compares a feedback condition with a non-feedback condition. Therapists in the feedback condition receive feedback after every fourth session. The feedback is given by two trained and independent raters. The raters are licenced and experienced psychotherapists. Therapists in the non-feedback condition receive no feedback during the psychotherapy.

ELIGIBILITY:
Therapists

Inclusion Criteria:

* Having successfully completed the interim audit
* Having started to treat ambulant patients
* Remaining at least 6 month in the ambulance

Exclusion Criteria:

-

Patients

Inclusion Criteria:

* Meeting ICD 10 criteria for a mental disorder
* Informed consent

Exclusion Criteria:

* Currently in psychotherapy
* Suicidal tendency
* Clinical diagnosis of alcohol or drug addiction, acute schizophrenia, schizoaffective disorder or bipolar disorder
* Clinical diagnosis of personality disorder cluster A (odd disorders) and B (dramatic, emotional or erratic)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Therapy Scale (CTS) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  external-assessment measure that assesses psychotherapeutic competency during a cognitive therapy session. CTS will be used by two trained raters licensed as psychological psychotherapists.

SECONDARY OUTCOMES:
Helping Alliance Questionaire (HAQ) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess therapeutic alliance from the therapists perspective (therapist version; HAQ-T) and the patients perspective (HAQ-P)
Berner Stundenbögen Version 2000 | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess therapeutic relationship from the therapists perspective (therapist version, TSTB) and the patients perspective (patient version; PSTB)
Global Assessment of Functioning (GAF) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  external measure to assess the global functioning of the patient
Supervisory Questionaire (SQ) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess the therapists self-opening
Supervisee Levels Questionaire (SLQ-R) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess the therapists self-awareness
Counseling Self-Estimate Inventory (COSE) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess self efficacy of the therapist
Fear of negative evaluation scale (Skala Angst vor negativer Bewertung; SANB) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess fear of evaluation
Brief Symptom Inventory (BSI) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess aspects of general psychopathology
Beck Depression Inventory II (BDI II) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess depressive symptoms
Beck Anxiety Inventory (BAI) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess anxiety symptoms
Client Satisfaction Questionaire (CSQ8) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess satisfaction with therapy
Health-related quality of life (SF-12) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Florian Weck, PhD, Principal Investigator — Goethe University
Locations (1):
- Department of Clinical Psychology and Psychotherapy of Goethe University, Frankfurt am Main, Hesse, Germany